CLINICAL TRIAL: NCT03217474
Title: A Randomized Controlled Clinical Trial of Corneal Debridement for the Treatment of Herpes Simplex Epithelial Keratitis
Brief Title: Femtosecond Laser-assisted Corneal Debridement for Herpes Simplex Keratitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chunxiao Wang (Other)
Responsible Party: Sponsor-Investigator, Chunxiao Wang, Clinical investigator, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017KYPJ052
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Herpes Simplex Keratitis
MeSH Terms: conditions — Keratitis, Herpetic | interventions — Ganciclovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FLDEB combined with GCV orally (Experimental): Femtosecond laser-assisted cornea debridement (FLDEB) combined with ganciclovir (GCV) orally.
  Interventions: Procedure: FLDEB; Drug: Ganciclovir (GCV); Device: Femtosecond laser
- GCV orally (Active Comparator): Ganciclovir (GCV) orally only
  Interventions: Drug: Ganciclovir (GCV)

INTERVENTIONS:
Procedure: FLDEB — The eye will be anesthetized, and femtosecond laser technology will be used to remove epithelial tissue (diameter: 8mm; depth: 100micron) that includes the loosened diseased corneal epithelial cells. Antibiotic ointments and drops will be instilled postoperatively.
  Other Names: Femtosecond laser-assisted corneal debridement
  Arms: FLDEB combined with GCV orally
Drug: Ganciclovir (GCV) — Patient will be treated with GCV orally (200mg, 3 times a day, for 14 days).
Device: Femtosecond laser — A commercial femtosecond laser to create a particular shaped graft for transplantation.
  Arms: FLDEB combined with GCV orally

SUMMARY:
The purpose of the study is to learn if adding femtosecond laser-assisted corneal debridement to a standard therapy of oral ganciclovir can help shorten the healing time of herpes simplex epithelial keratitis (HSK).

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 80 years old;
2. Epithelial ulceration in a dendritic or geographic pattern, characteristic of infection with herpes simplex virus, and within 7 days of onset;
3. Ulcer's stromal involvement < 120 micron, as indicated by anterior segment optical coherence tomography;
4. Informed consent signed by patient or legal guardian. Having the ability to comply with study assessments for the full duration of the study.

Exclusion Criteria:

1. Clinical signs of a cause other than herpes simplex virus for the epithelial keratitis;
2. Antivirus or corticosteroid treatment within 6 months;
3. Active stromal keratitis or iritis;
4. History of allergy or adverse reaction to ganciclovir;
5. High myopia with a spherical equivalent of -15.0 D or less;
6. Corneal or ocular surface infection within 30 days prior to study entry;
7. Ocular surface malignancy;
8. Uncontrolled diabetes with most recent Hemoglobin A1c greater than 8.5%;
9. Renal failure with creatinine clearance< 25ml/min;
10. Alanine aminotransferase > 40IU/L, or aspartate aminotransferase > 40IU/L;
11. Platelet levels < 150,000 or > 450,000 per microliter;
12. Hemoglobin < 12.0 g/dL (male) or < 11.0 g/dL (female);
13. Prothrombin time > 16s and activated partial thrombin time > 35s in patients not accepting anticoagulant therapy; An international normalized ratio greater than 3 in patients accepting anticoagulant therapy;
14. Pregnancy (positive test) or lactation;
15. Participation in another simultaneous medical investigation or clinical trial;
16. Severe cicatricial eye disease; Conjunctival scarring with fornix shortening;
17. Severe dry eye disease as determined by Schirmer's test < 2mm at least in one eye;
18. Any medical or social condition that in the judgement of the investigator would interfere with or serve as a contraindication to adherence to the study protocol or ability to give informed consent;
19. Active immunological diseases;
20. History of allo-limbal transplantation, penetrating keratoplasty or anti-glaucoma filtering surgeries.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Healing time | 14 ± 1 days
  Time to complete corneal epithelial healing

SECONDARY OUTCOMES:
Corneal re-epithelization | 14 ± 1 days
  Assessing complete corneal re-epithelization at day 14±1 using slit-lamp microcopy
Corneal opacity and vascularization | Baseline, 14 ± 1 days, 3 months
  Assessing corneal opacity and vascularization using slit-lamp microcopy
Best-corrected visual acuity | Baseline, 14 ± 1 days, 3 months
  Assessing best-corrected visual acuity using ETDRS chart
Corneal power and astigmatism | Baseline, 14 ± 1 days, 3 months
  Assessing changes of corneal power and astigmatism using autorefractor keratometer
Corneal sensation | Baseline, 14 ± 1 days, 3 months
  Assessing corneal sensation using Cochet-Bonnet esthesiometer
Recurrence | 3 months
  Assessing recurrent HSK using slit-lamp microcopy

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, M.D.Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Ting Huang, M.D.Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen Univerisity, Guangzhou, Guangdong, China